CLINICAL TRIAL: NCT01075919
Title: Cognitive and Mood Effects of DHA-rich and EPA-rich Fish Oil in Healthy Young Adults
Brief Title: Cognitive and Mood Effects of Docosahexaenoic Acid (DHA)-Rich and Eicosapentaenoic Acid (EPA)-Rich Fish Oil in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Ginsana SA (Other)
Responsible Party: Philippa Jackson, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16N1
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Cognitive Function; Mood
Keywords: n-3 PUFAs; Cognitive function; Healthy young adults; Fish oil; Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DHA-rich fish oil (Active Comparator): 1 g DHA-rich fish oil containing 450 mg DHA + 90 mg EPA
  Interventions: Dietary Supplement: n-3 PUFAs
- EPA-rich fish oil (Active Comparator): 1 g EPA-rich fish oil containing 300 mg EPA + 200 mg DHA
  Interventions: Dietary Supplement: n-3 PUFAs
- Placebo (Placebo Comparator): 1 g Olive oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-3 PUFAs — 1 g DHA-rich fish oil taken daily for 12 weeks
  Arms: DHA-rich fish oil
Dietary Supplement: Placebo — 1 g olive oil taken daily for 12 weeks
  Arms: Placebo
Dietary Supplement: n-3 PUFAs — 1 g EPA-rich fish oil taken daily for 12 weeks
  Arms: EPA-rich fish oil

SUMMARY:
To date, only a small handful of studies have assessed the effects of omega-3 polyunsaturated fatty acids (n-3 PUFAs) on cognitive function in healthy adults. The results from these studies are mixed, and have differed greatly in terms of methodology as regards sample size, treatment formulation and duration of the intervention. In order to address these issues, the present study aims to assess the effects of two different formulations of fish oil in parallel, and at doses consistent with the current recommended daily intake of oily fish, across a range of cognitive domains. The aim of the present investigation is therefore to specifically evaluate the effects of 12 weeks supplementation of DHA-rich fish oil and EPA-rich fish oil dietary supplements on cognitive function in healthy young adults maintaining a regular diet containing oily fish not more than once a week. Self-report mood assessments will form the secondary part of this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* 18-35 years
* Healthy
* No herbal supplements/prescription medications (excl. contraceptive pill)
* Non smoker
* Native English speaker

Exclusion Criteria:

* Consumes ≥ 1 portion oily fish/week
* takes omega-3 supplement
* Food allergies to treatment ingredients

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 12 weeks
  Performance is assessed using the COMPASS (Computerised Mental Performance Assessment) system, which presents a battery of standard cognitive tasks assessing aspects of attention, memory and executive function. The Cognitive Demand Battery (30 minutes)will also be administered and assesses cognitive performance under mental fatigue.

SECONDARY OUTCOMES:
Mood | 12 weeks
  Mood will be evaluated using Bond-Lader VAS and the Depression, Anxiety and Stress Scales.

CONTACTS AND LOCATIONS:
Overall Officials: Philippa A Jackson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- See also: Brain, Performance and Nutrition Research Centre, Northumbria University — http://www.nutrition-neuroscience.co.uk/